CLINICAL TRIAL: NCT03976115
Title: A Randomized, Double-Blind, Dose-escalating, Placebo Controlled, Phase I Study to Evaluate the Safety and Pharmacokinetics and Pharmacodynamics of DDO-3055 in Healthy Volunteers and Patients With Chronic Kidney Disease
Brief Title: A Study to Evaluate the Safety and Efficacy of DDO-3055 in Healthy Volunteers and Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: DDO-3055-101
Record Dates: First submitted 2019-05-29; First posted 2019-06-05 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. healthy volunteers (Experimental): 3x single dose of DDO-3055 and placebo
  Interventions: Drug: DDO-3055; Drug: Placebos
- 2. Patients with chronic kidney disease (Experimental): 3x single dose of DDO-3055 and placebo
  Interventions: Drug: DDO-3055; Drug: Placebos

INTERVENTIONS:
Drug: DDO-3055 — Oral
Drug: Placebos — Oral

SUMMARY:
This is a randomized, double-blind, dose-escalating, placebo controlled, Phase I study to evaluate the safety, pharmacokinetics and pharmacodynamics of DDO-3055 in healthy volunteers and patients with chronic kidney disease.

48 healthy volunteers will be enrolled in Part A, and 18 patients with chronic kidney disease will be enrolled in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:

Male or female volunteers aged 18 to 45 years of age inclusive ; Hemoglobin is 120 to 160 g/L; In good health, at the discretion of the investigator, as determined by: medical history, physical examination, vital sign assessment, 12-lead ECG, clinical laboratory evaluations.

- Patients with chronic kidney disease : Male or female patients with chronic kidney disease who are 18 to 45 years of age inclusive; Hemoglobin is ≤100 g/L; 30mL/min/1.73m2 ≤ eGFR ≤ 60mL/min/1.73m2（according to CKD-EPI formula）;

* Body weight is ≥ 50kg, and 19kg/m2 ≤ body mass index<26kg/m2 .
* Normal iron reserves (serum iron >61 g/dL and serum ferritin normal >30ng/mL).
* Signed informed consent.

Exclusion Criteria:

Healthy volunteers:

- The serum creatinine exceeded the upper limit of normal value in the screening period.

Healthy volunteers and patients with chronic kidney disease:

* Allergic to the study drug or any of its ingredients.
* Treating or treated with erythropoiesis stimulating agents for 1 month before screening.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or gamma-glutamyl transferase (GGT) or total bilirubin above 1.5 times normal upper limit (ULN) in the screening period.
* Have a history of blood donation or blood transfusion within 3 months.
* Vein blood collection is difficult or physical condition can not afford blood collection.
* Hepatitis b surface antigen (HBsAg), hepatitis c antibody (HCVAb), syphilis antibody, or human immunodeficiency virus (HIV) antibody test is positive in the screening period.
* Smoking 5 cigarettes per day on average within 3 months; or the average daily intake of alcohol within one week is more than 15g (15g alcohol is equivalent to 450mL beer or 150mL wine or 50mL low-alcohol liquor) or 2 days before taking the study drug and during the study period, tobacco, alcohol and caffeinated food or beverage are not prohibited, or those with special dietary requirements cannot comply with the unified diet.
* Those who have participated in clinical trials of any drug or medical device within 3 months prior to screening, or those who have participated in the drug trial within 5 half-lives prior to screening; any health product (within 1 week prior to administration), over-the-counter drug (2 weeks prior to administration) or prescription drug (1 month prior to administration) that affects the absorption, distribution, metabolism or excretion of the tested drug.
* With a history of drug abuse or positive screening/baseline test for substance abuse and drug urinalysis.
* During the study period and within 30 days after administration, men who are unwilling to take contraceptive measures and promise not to donate sperm are not allowed to participate in the study. Childbearing women who did not use contraception at least 14 days before administration; men and women who did not agree to use physical contraception during the study period.
* Women with serum HCG ≥ 5 mIU/mL or nursing in the screening period or baseline
* Any physical or mental illness or condition that may increase the risk of the study, affect the subject's compliance with the protocol, or affect the subject's ability to complete the study, as determined by the study physician.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Adverse Events(AEs) and Serious Adverse Events （SAEs） | from informed consent form signature to the end of the study (up to 14 days)
  Incidence of AEs and SAEs, incidence of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of DDO-3055 | Pre-dose to 72 hours after dose administration
Maximum observed serum concentration (Cmax) of DDO-3055 | Pre-dose to 72 hours after dose administration
Time to maximum observed serum concentration (tmax) of DDO-3055 | Pre-dose to 72 hours after dose administration
Time to elimination half-life (t1/2) of DDO-3055 | Pre-dose to 72 hours after dose administration
Apparent total clearance of the drug from plasma after oral administration (CL/F) of DDO-3055 | Pre-dose to 72 hours after dose administration
Apparent volume of distribution after non-intravenous administration (V/F) of DDO-3055 | Pre-dose to 72 hours after dose administration
Renal clearance of the drug from plasma (CLR) of DDO-3055 | Pre-dose to 72 hours after dose administration
Changes in red blood cell count relative to baseline | up to 14 days
Changes in reticulocyte count relative to baseline | up to 14 days
Changes in hemoglobin relative to baseline | up to 14 days
Changes in endogenous erythropoietin relative to baseline | up to 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China